CLINICAL TRIAL: NCT06349135
Title: Assessment of Serum Concentration of Interleukin-17 and Osteoprotegerin in Response to Surgical Trauma Induced by Management of Mandibular Fractures Via Intraoral Versus Extraoral Approaches: Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Aya Ayman Ahmed (Other)
Responsible Party: Sponsor-Investigator, Aya Ayman Ahmed, lecturer assistant, Cairo University
Organization: Cairo University (Other)
Other Study IDs: A.Ayman OMFS
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Management of Mandibular Fractures via Intraoral approach.: Management of Mandibular Fractures via Intraoral approach.
  Interventions: Procedure: Open Reduction & Internal Fixation
- Management of Mandibular Fractures via Extraoral approach.: Management of Mandibular Fractures via Extraoral approach.
  Interventions: Procedure: Open Reduction & Internal Fixation

INTERVENTIONS:
Procedure: Open Reduction & Internal Fixation — Open Reduction & Internal Fixation of Mandibular fracture either through intraoral or extraoral approaches.

SUMMARY:
Assessment of Serum Concentration of Interleukin-17 and Osteoprotegerin in Response to Surgical Trauma Induced by Management of Mandibular Fractures via Intraoral Versus Extraoral Approaches: Prospective Cohort Study

ELIGIBILITY:
Inclusion Criteria:

* Single mandibular fracture.
* ORIF is done by two plates fixation with titanium plates and screws.
* Age (18-50 years).
* Recent fracture (less than 2 weeks).

Exclusion Criteria:

* Pathological fractures.
* Medical compromised patient.
* Presence of concomitant injuries.
* Patients receive radiotherapy.
* Patients receive blood transfusion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with single mandibular fracture.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
IL-17 | 6- weeks
  Interleukin-17
OPG | 6- weeks
  Osteoprotegerin

SECONDARY OUTCOMES:
Blood Loss | in operation room
Operative time | Operative time in minutes